CLINICAL TRIAL: NCT00328484
Title: Exercise and Disability in COPD Patients
Brief Title: Comparison of Two Programs to Encourage Physical Activity in Individuals With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Michael J. Berry, PhD, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 387; R01HL053755-09 (NIH)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Exercise; Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Motor Activity; Emphysema; Bronchitis, Chronic | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Eleven month lifestyle activity program
  Interventions: Behavioral: Lifestyle Activity Program
- 2 (Active Comparator): Three month exercise program
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Lifestyle Activity Program — The lifestyle activity program will consist of 35 exercise and counseling sessions spaced over 11 months. This program will use cognitive-behavioral strategies to encourage physical activity at home. Participants will receive information on how to deal with COPD symptoms (including shortness of breath), goal-setting, social support, and motivation. Participants will also receive follow-up telephone calls from the program staff for additional support.
  Arms: 1
Behavioral: Exercise Program — The 3-month exercise program will consist of 36 1-hour exercise training sessions, conducted 3 times a week for 12 weeks.
  Arms: 2

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease. Symptoms include shortness of breath, wheezing, and difficulty exercising. Increasing exercise and physical activity may relieve the symptoms of COPD and may also slow the progression of the disease. The purpose of this study is to evaluate the effectiveness of a lifestyle activity program versus a traditional exercise program at increasing the amount of physical activity among individuals with COPD.

DETAILED DESCRIPTION:
COPD is a disease in which the lung airways are partly damaged and obstructed, making it difficult to breathe. It is the fourth leading cause of death in the United States. Cigarette smoking is the most common cause of COPD; however, breathing in other types of lung irritants, including pollution, dust, and chemicals, over a long period of time may also cause or contribute to COPD. The primary symptoms of COPD, exercise intolerance and shortness of breath, often result in physical activity limitations, which may lead to a decreased quality of life. While COPD is a chronic, incurable disease, individuals who incorporate exercise and physical activity into their daily lifestyle may reduce the symptoms and slow the progression of the disease. The purpose of this study is to compare the effectiveness of an overall lifestyle activity program versus a traditional exercise program on physical activity in individuals with COPD. The study will also evaluate the impact of the two programs on exercise capacity, physical function, self-reported disability, and health-related quality of life.

Participants with COPD will be randomly assigned to either an 11-month lifestyle activity program or a traditional 3-month exercise program. The lifestyle activity program will consist of 35 exercise and counseling sessions spaced over 11 months. This program will use cognitive-behavioral strategies to encourage physical activity at home. Participants will receive information on how to deal with COPD symptoms (including shortness of breath), goal-setting, social support, and motivation. Participants will also receive follow-up telephone calls from the program staff for additional support. The 3-month exercise program will consist of 36 1-hour exercise training sessions, conducted 3 times a week for 12 weeks.

All participants will attend 4 baseline study visits at which their medical history will be reviewed and standardized questionnaires will be completed to assess mood, depression, social factors, COPD symptoms, and physical activity levels. Participants will undergo a physical examination; a blood draw for laboratory testing; and spirometry, lung function, exercise, and strength tests. These measures will be assessed again at 3, 6, and 12 months; the 3- and 12-month assessments will occur over four study visits, and the 6-month assessment will occur over two study visits.

ELIGIBILITY:
Inclusion Criteria:

* Expiratory airflow limitation such that FEV1/FVC is less than or equal to 70% and the FEV₁ is greater than or equal to 20% of the predicted amount
* Physical disability, including self-reported difficulty with walking a city block, climbing stairs, lifting and carrying groceries, performing household activities such as cleaning and doing yard work, or getting out of a chair
* Currently lives within a 35-mile radius of Wake Forest University
* Plans to reside in Forsyth County, North Carolina for the entire study
* Willing and able to participate in all aspects of the trial

Exclusion Criteria:

* Undergoing treatment for cancer
* Severe congestive heart failure
* Stroke
* Peripheral vascular disease
* Coronary artery disease
* Valvular heart disease
* Major psychiatric disease
* Severe anemia
* Liver or kidney disease
* Uncontrolled diabetes or hypertension
* Orthopedic impairment
* Blindness or deafness
* Oxygen desaturation during exercise to less than 90%, at a heart rate less than 50% of predicted maximum for participant's age and without supplemental oxygen
* Inability to exercise due to a physical disability or positive exercise stress test
* Alcohol consumption of greater than two drinks per day in the 2 months prior to study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2002-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Amount of time engaged in moderate physical activity each week | Measured at Year 1

SECONDARY OUTCOMES:
Health related quality of life | Measured at Year 1
Self-reported disability | Measured at Year 1
Physical function | Measured at Year 1
Exercise capacity | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Berry, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Foy CG, Wickley KL, Adair N, Lang W, Miller ME, Rejeski WJ, Woodard CM, Berry MJ. The Reconditioning Exercise and Chronic Obstructive Pulmonary Disease Trial II (REACT II): rationale and study design for a clinical trial of physical activity among individuals with chronic obstructive pulmonary disease. Contemp Clin Trials. 2006 Apr;27(2):135-46. doi: 10.1016/j.cct.2005.11.011. Epub 2006 Feb 2. PMID 16458075
- [Background] Katula JA, Rejeski WJ, Wickley KL, Berry MJ. Perceived difficulty, importance, and satisfaction with physical function in COPD patients. Health Qual Life Outcomes. 2004 Mar 31;2:18. doi: 10.1186/1477-7525-2-18. PMID 15056389
- [Background] Berry MJ, Adair NE, Rejeski WJ. Use of peak oxygen consumption in predicting physical function and quality of life in COPD patients. Chest. 2006 Jun;129(6):1516-22. doi: 10.1378/chest.129.6.1516. PMID 16778269
- [Derived] Berry MJ, Rejeski WJ, Miller ME, Adair NE, Lang W, Foy CG, Katula JA. A lifestyle activity intervention in patients with chronic obstructive pulmonary disease. Respir Med. 2010 Jun;104(6):829-39. doi: 10.1016/j.rmed.2010.02.015. Epub 2010 Mar 26. PMID 20347286